CLINICAL TRIAL: NCT00163267
Title: Follow-up Management of Peripheral Arterial Intervention With Clopidogrel MIRROR-Study
Brief Title: Mirror Trial - Follow-Up Management of Peripheral Arterial Intervention With Clopidogrel
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Mirror Trial, University of Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: mi-1; D.3100340
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2007-04

CONDITIONS: Peripheral Vascular Diseases
Keywords: peripheral arterial intervention; atherosclerosis; platelets; Age above 18
MeSH Terms: conditions — Peripheral Vascular Diseases; Atherosclerosis | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- ASS + Placebo (Placebo Comparator): control arm
  Interventions: Drug: clopidogrel
- ASS + Plavix (Active Comparator): active drug
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: clopidogrel — Best endovascular treatment either with one or the other drug arm should be investigated

SUMMARY:
The Mirror Study is a randomized, double-blinded mono-centre trial the access the periinterventinal and postinterventional administration of clopidogrel in patients with peripheral vascular disease.

DETAILED DESCRIPTION:
Clopidogrel is approved for secondary prevention of atherosclerosis in patients with peripheral vascular disease. Currently there are no data about the amount of platelet activation during peripheral arterial intervention, the effect of clopidogrel on platelet adhesion and its clinical impact.

Patients with chronic peripheral arterial disease receive placebo or clopidogrel before the intervention and for 6 months in follow-up. Platelet activation, the effect on macro-and microcirculation will be assessed as well as clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral arterial disease which requires intervention

Exclusion Criteria:

* Patient already on coumadin or clopidogrel
* Acute onset of PVD symptoms
* Patient requiring an operation
* Contraindication to aspirin and clopidogrel

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Platelet activation during and after the intervention | 6-12 hours
  measured in a chandler loop model

SECONDARY OUTCOMES:
ABI | before patients leaves the hospital and at 6 months
  as treatment effect
clinical improvement | up to 6 months
  dependent on the additional drug treatment
Safety | up to 6 months
  dependent on the drug treatment with the endovascular treatment
rate of occlusions | wihtin 6 months
  dependent on drug treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Tepe, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital of Tuebingen, Tübingen, Germany

REFERENCES:
- [Derived] Strobl FF, Brechtel K, Schmehl J, Zeller T, Reiser MF, Claussen CD, Tepe G. Twelve-month results of a randomized trial comparing mono with dual antiplatelet therapy in endovascularly treated patients with peripheral artery disease. J Endovasc Ther. 2013 Oct;20(5):699-706. doi: 10.1583/13-4275MR.1. PMID 24093324